CLINICAL TRIAL: NCT04542239
Title: Inclined Positioning and Infant Gastroesophageal Reflux Indicators
Brief Title: Inclined Positioning and Infant Gastroesophageal Reflux
Acronym: Infant GER
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Iron Mountains (Unknown)
Responsible Party: Principal Investigator, Ian M. Paul, MD, Professor of Pediatrics, Milton S. Hershey Medical Center
Other Study IDs: HRP591
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with GER: Infants (N=25) meeting inclusion/exclusion criteria
- Controls without GER: Infants (N=10) meeting inclusion/exclusion criteria, but no GER

SUMMARY:
The purpose of this voluntary research study is to evaluate the extent to which infants with Gastroesophageal Reflux (GER) exhibit oxygen desaturation (low oxygen levels in their blood) and bradycardia (slow heart rate) in supine (lying flat on back) and inclined positions.

DETAILED DESCRIPTION:
Mothers will bring their infants to the Clinical Research Center where they will be escorted to a private room. Participants will proceed to feed their infant a typical liquid meal (i.e. breastmilk or formula). Within 15 minutes of completion of the feed, infants will be placed in the prototype infant reclining device at either 0, 10, 18, or 28 degrees of incline. Infants will spend 15 minutes at each level of incline in a randomly assigned order. During this time period that each infant is under observation the infant may be entertained/distracted/comforted with white noise, music or other forms of distraction as determined by the mother or study team. Mothers may touch/caress their infant or use a pacifier to soothe infant as needed so long as each 15 minute segment is completed. Following each 15 minute segment, a "washout" period will be used such that the next 15 minute segment will not begin for a minimum of 1 minute to a maximum of 5 minutes in duration before the next incline position is begun. This allows for a clean start and stop period for each 15 minute segment that is not impacted by either the prior position or the change to the new position. This also allows mothers or study staff to pick up and comfort the infant.

During each of the four 15 minute segments, infants will be monitored using the Masimo RAD-97 pulse oximeter with data continuously collected regarding oxygen saturation and heart rate in 2-second intervals. The oxygen saturation probe will preferably be attached to a big toe, but can be placed in alternative spots consistent with usual clinical care such that a consistent reading of heart rate and oxygen saturation are recorded. A study coordinator will complete a data collection form for each segment characterizing whether GER occurred (spit-up into mouth or outside of mouth), the number of GER episodes as well as a subjective assessment of degree crying/fussing, hiccups, back arching, and breathing difficulty. The coordinator will also have a timer to measure the duration of crying in each position. Infants will be video recorded as a backup method for symptom assessment and for qualitative assessments by the study sponsor.

ELIGIBILITY:
Inclusion Criteria:

* born at >= 34 weeks gestation
* weight for age >= 10th percentile
* No serious medical conditions
* English-speaking parent capable of consenting
* Diagnosis of GER from healthcare provider (not necessary for controls)
* 4 or more visible spit-ups (mouth or nose) per day for at least 5 days OR 2 or more spit-ups out of the nose per day for at least 5 days OR I-GERQ score >=16 (not necessary for controls)
* If applicable, parent willing to refrain from giving medication for GER for 12 hours prior to study participation

Exclusion Criteria:

* Signs of a more serious or complex illness including weight loss, lethargy, fever, excessive irritability/pain, bulging fontanelle, seizures, macro/microcephaly, bilious vomiting, hematemesis, chronic diarrhea, rectal bleeding, suspicions of GI obstruction
* History of a Brief Resolved Unexplained Event (BRUE)
* Use of a Home Apnea Monitor prescribed by a healthcare provider

Ages: 1 Month to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be identified through providers in the Divisions of Academic General Pediatrics, Hospital Pediatrics, and Pediatric Gastroenterology. The Department of Family and Community Medicine may also refer participants to the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Number of hypoxic episodes | 1 hour observation period
  Evaluate the extent to which infants exhibit oxygen desaturation (oxygen saturation <94%) in each position
Number of bradycardia episodes | 1 hour observation period
  Evaluate the extent to which infants exhibit bradycardia (heart rate <100 beats per minute) in each position
Number of observed regurgitations | 1 hour observation periods
  Evaluate the extent to which infants exhibit clinical signs and symptoms of post-feed regurgitation in each position

SECONDARY OUTCOMES:
Time spent in hypoxic episodes | 1 hour observation period
  Minutes spent in hypoxia in each position
Time spent in bradycardic episodes | 1 hour observation period
  Minutes spent in bradycardia in each position
Time spent fussing or crying | 1 hour observation period
  Minutes spent fussing or crying in each position
Observed cyanosis episodes | 1 hour observation period
  Number of episodes of observed cyanosis (turning blue) in each position
Subjective assessment of crying, hiccups, back arching, and respiratory distress | 1 hour observation period
  Yes/no answer in each position
Subjective maternal perception of infant comfort in each position | 1 hour observation period
  very comfortable, comfortable, neither comfortable nor uncomfortable, uncomfortable, very uncomfortable

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Paul IM, Shedlock KE, Schaefer EW, Stoute EJ, Rosen R. Pilot Study of Inclined Position and Infant Gastroesophageal Reflux Indicators. JPGN Rep. 2023 Apr 24;4(2):e312. doi: 10.1097/PG9.0000000000000312. eCollection 2023 May. PMID 37200720